CLINICAL TRIAL: NCT03523897
Title: A Prospective Study to Examine Patient Satisfaction, Function, and Limb Alignment Outcomes for Mako Versus Non-Mako Total Knee Replacements
Brief Title: A Prospective Study to Evaluate Robot Assisted Total Knee Replacement Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient research coordinating support to continue recruitment and data collection
Sponsor: Virtua Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VirtuaHealth-Mako
Record Dates: First submitted 2018-03-13; First posted 2018-05-14 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Primary Osteoarthritis of Knee Nos

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Robot Assisted Total Knee Replacement (Active Comparator): In addition to expert judgment and hand-eye coordination, the surgeon also relies on a robot in making cuts within the pre-determined diseased areas of the joints and placing the implants. This is made possible by uploading 3-dimensional (3D) images of the knee joints into the robot prior to surgery. The robot uses these 3D images to guide the surgeon during the procedure. The 3D images are obtained from a computerized tomography (CT) scan that combines a series of X-ray images taken from different angles to create cross-sectional images of the bones.
  Interventions: Procedure: Robot Assisted Total Knee Replacement
- Traditional Total Knee Replacement (Active Comparator): The traditional method where the surgeon employs mechanical guides, expert judgment, and natural hand-eye coordination in making the necessary cuts to prepare the bone for the implant as well as in placing the implant.
  Interventions: Procedure: Traditional Total Knee Replacement

INTERVENTIONS:
Procedure: Robot Assisted Total Knee Replacement — A robotic-assisted surgical procedure to treat a condition in which the patient's knee joints become diseased or injured due to a loss of cartilage that acts as a protective cushion between the knee joints
  Arms: Robot Assisted Total Knee Replacement
Procedure: Traditional Total Knee Replacement — A surgical procedure using mechanical guides to treat a condition in which the patient's knee joints become diseased or injured due to a loss of cartilage that acts as a protective cushion between the knee joints
  Arms: Traditional Total Knee Replacement

SUMMARY:
This study aims to see if outcomes for patients that receive the traditional total knee replacement surgical technique are different than the outcomes for patients that receive robot-assisted total knee replacement. The outcomes we will be tracking include:

1. Patients' self-reported awareness of their artificial joints during activities of daily living;
2. Patient's self-reported pain, other symptoms, function in daily living, function in sport and recreation, and knee-related quality of life;
3. Patients' self-reported general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning and mental health;
4. The accuracy of implant placement and limb alignment

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Diagnosed with primary osteoarthritis and cleared to undergo total knee arthroplasty at the Virtua JRI
3. Willing to provide informed consent, participate in study, and comply with study protocol

Exclusion Criteria:

1. Pregnant or contemplating pregnancy prior to surgery;
2. Worker's compensation or personal injury related to knee (clinical outcomes have been shown to be less predictable and often poorer in this patient group; there may also exist potential issues with reimbursement)
3. Post-traumatic arthropathy (clinical outcomes have been shown to be less predictable; pre-operative deformity and risk factors are greater and difficult to propensity-match between groups)
4. Self-pay patients or patients whose insurance are known to typically decline reimbursement for preoperative CT scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Reid, MD, Principal Investigator — Virtua Joint Replacement Institute
Locations (1):
- Virtua Joint Replacement Institute, Voorhees Township, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Plan to pblish study outcomes in a relevant orthopedic journal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robot Assisted Total Knee Replacement | Traditional Total Knee Replacement
Started | 39 | 53
Completed | 0 | 0
Not Completed | 39 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robot Assisted Total Knee Replacement | Traditional Total Knee Replacement | Total
Number analyzed (Participants) | 39 | 53 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 38 | 53 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 59
  Male | 13 | 20 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 38 | 51 | 89
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 53 | 92

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Forgotten Joint Score (FJS)
Description: The FJS is a self-completed 12-item questionnaire used to assess patients' awareness of their artificial joint during activities of daily living on an awareness scale of 0 (never) to 4 (mostly)
Time Frame: 1 year
Population: Study canceled due to lack of resources. The personnel responsible for collecting data left the hospital system before any data was collected and the investigators involved did not have the time necessary to collect and organize data. Therefore, no data was collected at the 1-year timeframe, leading to no data available for analysis.
Arm/Group | Robot Assisted Total Knee Replacement | Traditional Total Knee Replacement
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Reported Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS is a knee-specific instrument used to evaluate short-term and long-term symptoms and function in subjects with knee injury and osteoarthritis. It consists of 42 questions in 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Robot Assisted Total Knee Replacement | Traditional Total Knee Replacement
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient Reported Veterans Rand 12-item Health Survey Score (VR-12)
Description: The VR-12 is a 12-item questionnaire corresponding to eight principal physical and mental health domains including general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning and mental health.
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: The Mechanical Alignment of the Post-operative Limb
Description: The mechanical alignment of the entire post-operative limb will be measured at 6 weeks by long-limb radiograph cassettes and compared to the pre-operative plan for accuracy and deviation less than or greater than 3 degrees from the intended target. From each treatment group, the percentage of patients with radiographic outliers (deviation greater that 3 degrees from the expected implant placement) will be compared.
Time Frame: 6 weeks postoperatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data was not collected
Description: Data was not collected
Arm/Group | Robot Assisted Total Knee Replacement | Traditional Total Knee Replacement
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT03523897/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT03523897/ICF_001.pdf